CLINICAL TRIAL: NCT05864534
Title: A Phase 2a Trial of Immune Modulation in Combination With Ultrasound-mediated Blood Brain Barrier Opening in Patients With Newly Diagnosed Glioblastoma
Brief Title: Phase 2a Immune Modulation With Ultrasound for Newly Diagnosed Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agenus Inc. (Industry); CarThera (Industry)
Responsible Party: Principal Investigator, Adam M Sonabend, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU23C03
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Newly Diagnosed Glioblastoma; Glioblastoma, Isocitric Dehydrogenase (IDH)-Wildtype; Gliosarcoma; Glioblastoma Multiforme
Keywords: Immunotherapy; Ultrasound; Blood-brain barrier; Sonocloud; Balstilimab (BAL); Botensilimab (BOT); Doxorubicin (DOX)
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — balstilimab; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Blood-brain barrier opening with concomitant BAL, BOT, DOX (Experimental): Patients will undergo implantation of Sonocloud-9 after completion of radiotherapy. Within 21 days after implant, ultrasound-based BBB opening with concomitant administration of DOX (30 mg) + BAL (450 mg) every 3 weeks, and BOT (dose 1mg/kg) every 6 weeks will be initiated.
  Interventions: Drug: Balstilimab; Drug: Botensilimab; Drug: Liposomal Doxorubicin; Device: Sonocloud-9 (SC-9)

INTERVENTIONS:
Drug: Balstilimab — Balstilimab 450 mg IV over 30 minutes every 3 weeks
  Other Names: BAL
Drug: Botensilimab — Botensilimab1mg/kg mg IV over 30 minutes every 6 weeks
  Other Names: BOT
Drug: Liposomal Doxorubicin — Liposomal Doxorubicin 30 mg IV over 30 minutes every 3 weeks
  Other Names: DOX
Device: Sonocloud-9 (SC-9) — Device activation of 9 ultrasound emitters during IV injection of microbubbles every 3 weeks
  Other Names: SC-9

SUMMARY:
Brain tumor treatment is hampered by the blood-brain barrier (BBB). This barrier prevents drugs carried in the bloodstream from getting into the brain. If the BBB can be opened, making it temporarily more permeable, drugs may able to better reach the brain tumor. In this trial we will implant a novel device with 9 ultrasound emitters, allowing temporary and reversible opening of the BBB to maximize brain penetration of drugs that modulate the immune system. The device will be implanted after radiation is completed. Immune modulating drugs will be given every 3 weeks in conjunction with activation of the device to open the BBB.

The objectives of this trial are to establish whether it is safe and feasible to administer immune modulating drugs in this manner, and identify whether the treatment is effective in treating glioblastoma.

DETAILED DESCRIPTION:
Eligible patients will undergo implant of the Soncloud-9 device within 1-5 weeks of completion of radiotherapy. About 1-3 weeks after surgery, patients will undergo sonication and intravenous administration of balstilimab, botensilimab and liposomal doxorubicin. Brain MRI will be done to quantify extent of blood brain barrier opening. The dose for balstilimab is 450 mg every 3 weeks. The dose for botensilimab is 1mg/kg every 6 weeks. The dose for liposomal doxorubicin is 30 mg every 3 weeks. Sonication and administration of study agents will continue every 3 weeks (21 days= 1 cycle) for a total of 9 cycles (approx. 6 months). Additional cycles may be considered if deemed beneficial and in the patient's best interest. Blood samples for circulating tumor DNA will also be collected before and after each sonication. The first 6 patients will comprise a safety run-in cohort with intensified safety monitoring through the end of the second cycle.

ELIGIBILITY:
Inclusion Criteria:

* Have newly diagnosed pathologically proven glioblastoma, isocitric dehydrogenase-1/2 wild-type
* Tumor with methyl guanine methyl transferase (MGMT) gene promoter unmethylated
* Available paraffin embedded tumor tissue for the study
* Have completed standard radiotherapy with or without temozolomide
* 18 years of age or older
* Able to undergo contrast-enhanced MRI
* Have an Eastern Cooperative Oncology Group/World Health Organization performance status ≤ 2
* Size and location of the residual tumor and/or resection cavity must allow to be able to be covered by the sonication field
* Have not received any prior treatment with immunotherapeutic agents treatments for glioblastoma or other indications
* Have the ability to understand and willingness to sign a written informed consent prior to registration on study.
* Be willing and able to comply with the protocol.
* Have adequate organ and bone marrow function
* Agree to use adequate contraception if appropriate

Exclusion Criteria: Patients will be ineligible if they have:

* Multifocal tumor (unless all localized in a 50-mm diameter area accessible to ultrasound field) or tumor located in the posterior fossa.
* Uncontrolled epilepsy.
* Received other investigational agents within 2 weeks of registration
* Received prior therapy with or have history of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in this study.
* Contraindication to checkpoint inhibitor therapy (e.g., history of autoimmune disease)
* Uncontrolled illness
* History of active malignancy other than the brain tumor within 12 months prior to registration.
* Are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Unacceptable toxicity rate | 42 days
  Unacceptable toxicity rate in cycle 1 of < 33%
Landmark survival analyses | 18 months
  Overall survival and progression-free survival at 12 and 18 months, as well as median progression-free and overall survival.

SECONDARY OUTCOMES:
Predictive value of phospho-extracellular signal-related kinase (p-ERK) expression | 18 months
  Predictive value of baseline tissue p-ERK expression for response/benefit of immunotherapy
Response rate | 18 months
  Measurement of tumor shrinkage using Response Assessment in Neuro-oncology criteria in those with residual or tumor

OTHER OUTCOMES:
Patterns of recurrence | 18 months
  Patterns of recurrence by magnetic resonance imaging related to sonication field
Immune profile | 12 months
  Analysis of nucleic acid/exosomes and peripheral blood cell for correlation with progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Adam Sonabend, MD, Principal Investigator — Northwestern University; Roger Stupp, MD, Study Director — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Das R, Verma R, Sznol M, Boddupalli CS, Gettinger SN, Kluger H, Callahan M, Wolchok JD, Halaban R, Dhodapkar MV, Dhodapkar KM. Combination therapy with anti-CTLA-4 and anti-PD-1 leads to distinct immunologic changes in vivo. J Immunol. 2015 Feb 1;194(3):950-9. doi: 10.4049/jimmunol.1401686. Epub 2014 Dec 24. PMID 25539810
- [Background] O'Malley DM, Oaknin A, Monk BJ, Selle F, Rojas C, Gladieff L, Berton D, Leary A, Moore KN, Estevez-Diz MDP, Hardy-Bessard AC, Alexandre J, Opperman CP, de Azevedo CRAS, Randall LM, Feliu WO, Ancukiewicz M, Ray-Coquard I. Phase II study of the safety and efficacy of the anti-PD-1 antibody balstilimab in patients with recurrent and/or metastatic cervical cancer. Gynecol Oncol. 2021 Nov;163(2):274-280. doi: 10.1016/j.ygyno.2021.08.018. Epub 2021 Aug 25. PMID 34452745
- [Background] Treat LH, McDannold N, Zhang Y, Vykhodtseva N, Hynynen K. Improved anti-tumor effect of liposomal doxorubicin after targeted blood-brain barrier disruption by MRI-guided focused ultrasound in rat glioma. Ultrasound Med Biol. 2012 Oct;38(10):1716-25. doi: 10.1016/j.ultrasmedbio.2012.04.015. Epub 2012 Jul 19. PMID 22818878
- [Background] Beccaria K, Sabbagh A, de Groot J, Canney M, Carpentier A, Heimberger AB. Blood-brain barrier opening with low intensity pulsed ultrasound for immune modulation and immune therapeutic delivery to CNS tumors. J Neurooncol. 2021 Jan;151(1):65-73. doi: 10.1007/s11060-020-03425-8. Epub 2020 Feb 28. PMID 32112296
- [Background] Duerinck J, Schwarze JK, Awada G, Tijtgat J, Vaeyens F, Bertels C, Geens W, Klein S, Seynaeve L, Cras L, D'Haene N, Michotte A, Caljon B, Salmon I, Bruneau M, Kockx M, Van Dooren S, Vanbinst AM, Everaert H, Forsyth R, Neyns B. Intracerebral administration of CTLA-4 and PD-1 immune checkpoint blocking monoclonal antibodies in patients with recurrent glioblastoma: a phase I clinical trial. J Immunother Cancer. 2021 Jun;9(6):e002296. doi: 10.1136/jitc-2020-002296. PMID 34168003
- [Background] Shimozaki K, Sukawa Y, Sato Y, Horie S, Chida A, Tsugaru K, Togasaki K, Kawasaki K, Hirata K, Hayashi H, Hamamoto Y, Kanai T. Analysis of risk factors for immune-related adverse events in various solid tumors using real-world data. Future Oncol. 2021 Jul;17(20):2593-2603. doi: 10.2217/fon-2020-0861. Epub 2021 Apr 21. PMID 33878916
- [Derived] Kim KS, Habashy K, Gould A, Zhao J, Najem H, Amidei C, Saganty R, Arrieta VA, Dmello C, Chen L, Zhang DY, Castro B, Billingham L, Levey D, Huber O, Marques M, Savitsky DA, Morin BM, Muzzio M, Canney M, Horbinski C, Zhang P, Miska J, Padney S, Zhang B, Rabadan R, Phillips JJ, Butowski N, Heimberger AB, Hu J, Stupp R, Chand D, Lee-Chang C, Sonabend AM. Fc-enhanced anti-CTLA-4, anti-PD-1, doxorubicin, and ultrasound-mediated blood-brain barrier opening: A novel combinatorial immunotherapy regimen for gliomas. Neuro Oncol. 2024 Nov 4;26(11):2044-2060. doi: 10.1093/neuonc/noae135. PMID 39028616